CLINICAL TRIAL: NCT06090331
Title: An Expanded Access Program for the Non-invasive Detection of Clear Cell Renal Cell Carcinoma (ccRCC) in Patients With Renal Masses Utilizing 89Zirconium-labelled Girentuximab (89Zr-DFO-girentuximab)
Brief Title: 89Zr-DFO-girentuximab Expanded Access Program (EAP)
Status: Available | Type: Expanded Access
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 89Zr-TLX250-007
Record Dates: First submitted 2023-10-12; First posted 2023-10-19 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: clear cell renal cell carcinoma; PET/CT imaging; 89Zr-girentuximab
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Diagnostic Test: 89Zr-DFO-girentuximab — Single IV administration on Day 0, followed by diagnostic scan on Day 5 +/- 2 days.

SUMMARY:
The purpose of this Expanded Access Program (EAP) is to enable the use of 89Zr-DFO-girentuximab with positron emission tomography/computed tomography (PET/CT) imaging to non-invasively detect carbonic anhydrase 9 (CAIX)-expressing clear cell renal cell carcinoma (ccRCC) in patients with renal masses as determined by conventional imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Written and voluntarily given informed consent.
2. Male or female ≥ 18 years of age.
3. Imaging evidence of renal mass(es) obtained from conventional diagnostic imaging with CT or MRI (without and with contrast enhancement) based on national standards that is not older than 90 days on Day 0, and that was performed before any screening procedure.
4. Negative urine/serum pregnancy tests in female patients of childbearing potential.
5. Consent to practice highly effective contraception until a minimum of 42 days after IV 89Zr-DFO-girentuximab administration.

Exclusion Criteria:

1. Renal mass known to be a metastasis of another primary tumor.
2. Active non-renal malignancy requiring therapy during and up to EOT visit.
3. Radiotherapy or immunotherapy within 4 weeks (28 days) prior to the planned administration of 89Zr-DFO-girentuximab or continuing adverse effects (> grade 1 using Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) from such therapy.
4. Planned antineoplastic therapies (for the period between IV administration of 89Zr-DFO-girentuximab and imaging).
5. Previous administration of any radionuclide within 10 of its half-lives before Day 0.
6. Serious non-malignant disease (e.g., psychiatric, infectious, autoimmune, or metabolic), that may interfere with the objectives of the program or with the safety or compliance of the subject, as judged by the Investigator.
7. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the program.
8. Exposure to any experimental diagnostic or therapeutic drug within 30 days from the date of planned administration of 89Zr-DFO-girentuximab.
9. Women who are pregnant or breastfeeding.
10. Known hypersensitivity to girentuximab or DFO (desferoxamine).

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Arkansas Urology, Little Rock, Arkansas
  - UCLA, Los Angeles, California
  - University of Florida College of Medicine Jacksonville, Jacksonville, Florida
  - Biogenix Molecular, Miami, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Indiana University, Bloomington, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Munson Medical Center, Traverse City, Michigan
  - Xcancer, Omaha, Nebraska
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Kettering Health Main Campus, Kettering, Ohio
  - Urology Associates, PC, Nashville, Tennessee
  - Austin Radiological Association, Austin, Texas
  - UT Southwestern, Dallas, Texas
  - Urology San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah